CLINICAL TRIAL: NCT07048210
Title: Investigation of the Relationship Between Diaphragm Muscle Function and Urinary Incontinence in Stroke Patients
Brief Title: Diaphragm Function and Urinary Incontinence in Stroke
Status: Not yet recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Other Study IDs: IstinyeUni-STROKE-2025
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Stroke
Keywords: Diaphragm; Urinary Incontinence; Stroke; Respiratory Function
MeSH Terms: conditions — Stroke; Urinary Incontinence; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke Patients: 50 individuals diagnosed with stroke will undergo assessments of diaphragmatic function, respiratory muscle strength and endurance, and urinary incontinence.

SUMMARY:
Stroke affects respiratory functions by causing structural and strength impairments in both inspiratory and expiratory respiratory muscles. Weakening of the diaphragm leads to a decrease in maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP), which may result in respiratory insufficiency, postural instability, and urinary incontinence (UI). Additionally, post-stroke reduction in diaphragmatic mobility and decreased activity of the diaphragm and abdominal muscles on the paretic side may disrupt the piston mechanism between the diaphragm and pelvic floor muscles. These mechanical changes may trigger the development of urinary incontinence. This study aims to investigate the relationship between diaphragm muscle strength and endurance and urinary incontinence in 50 stroke patients. In addition, diaphragmatic function and posture-related respiratory changes will be evaluated using functional tests based on the Dynamic Neuromuscular Stabilization (DNS) approach. The relationship between respiratory muscle strength (MIP, MEP) and endurance and the scores of the Urogenital Distress Inventory (UDI-6) and the Incontinence Impact Questionnaire (IIQ-7) will be analyzed. Furthermore, individuals with and without urinary incontinence symptoms will be evaluated in terms of diaphragmatic function and contribution to respiration.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40 and 75 years,
* Diagnosed with hemorrhagic or ischemic stroke confirmed by computed tomography (CT) or magnetic resonance imaging (MRI) conducted by a specialist physician,
* Presence of urinary incontinence,
* No other orthopedic, rheumatologic, or neurological diagnoses apart from stroke,
* Ability to understand the investigator's instructions and a score of ≥24 on the Mini-Mental State Examination (MMSE),
* Voluntary participation in the study,
* Ability to speak and understand Turkish.

Exclusion Criteria:

* Presence of serious diseases affecting vital organs such as the heart, lungs, liver, or kidneys,
* Presence of a genitourinary infection,
* Pelvic organ prolapse at stage 3 or higher,
* Uncontrolled cardiopulmonary or unstable chronic diseases,
* Presence of one or more neurological disorders that may cause balance impairments,
* Severe cognitive, speech, or visual impairments,
* History of urogynecological surgery within the past 6 months,
* History of abdominal surgery within the past 6 months.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bahçelievler Medical Park Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2025-08-25 (Estimated); Study Completion 2025-09-29 (Estimated)

PRIMARY OUTCOMES:
Diaphragm Muscle Function | Baseline (single assessment)
  Diaphragm muscle function will be assessed using the Dynamic Neuromuscular Stabilization (DNS) approach. The evaluation consists of three components: (1) the diaphragm's contribution to respiration, (2) its role in postural stabilization, and (3) active respiration during postural stabilization. Each component will be rated separately using a 4-point scale: none (3), mild (2), moderate (1), and severe (0). Higher total scores reflect greater impairment in diaphragm-related respiratory function.
Urogenital Distress Inventory (UDI-6) | Baseline (single assessment)
  The Urogenital Distress Inventory (UDI-6) consists of 6 items and is rated on a four-point Likert scale. The total score ranges from 0 to 18, with higher scores indicating greater symptom distress and a more impaired quality of life.
Incontinence Impact Questionnaire (IIQ-7) | Baseline (single assessment)
  The Incontinence Impact Questionnaire (IIQ-7) consists of 7 items and is rated on a four-point Likert scale. The total score ranges from 0 to 21, with lower scores indicating less impact on quality of life.

SECONDARY OUTCOMES:
Respiratory Muscle Strength | Baseline (single assessment)
  Respiratory muscle strength will be assessed using a portable device capable of measuring maximal inspiratory (MIP) and expiratory (MEP) mouth pressures electronically (MicroRPM, Micro Medical, Kent, UK). Measurements will be conducted with the participant in a seated position, wearing a nose clip to prevent air leakage. For MIP, the participant will perform a maximal exhalation followed by a maximal inhalation against an occluded airway for at least 1.5 seconds. For MEP, a maximal inhalation will be followed by a maximal exhalation under the same conditions. Each measurement will be repeated three times with less than 10% variability, and the highest value will be used for analysis.
Respiratory Muscle Endurance | Baseline (single assessment)
  Respiratory muscle endurance will be assessed using a threshold loading test with the PowerBreathe device (HaB International Ltd., Southam, UK). The test will begin at 20% of the participant's maximal inspiratory pressure (MIP) and will be increased in two-minute intervals to 40%, 60%, 80%, and finally 100% of MIP. During the test, the device will be placed in the participant's mouth and a nose clip will be used to prevent nasal breathing. Participants will be instructed to breathe through the mouth for 10 minutes. Oxygen saturation and perceived dyspnea will be measured before the test, at the end of each two-minute stage, and after the test. Test results will be calculated by multiplying the total test duration by the corresponding pressure level at each stage.

IPD SHARING:
Plan to Share IPD: Yes
The study will share de-identified, summary-level outcome data, including group-level means, standard deviations, effect sizes, and p-values derived from statistical analyses. These data will be provided to support transparency and allow for interpretation of the study findings.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Summary-level data and supporting documents (e.g., study protocol and statistical analysis plan) will be available within 12 months following the final publication of study results and will remain accessible for at least 5 years via institutional repository or upon reasonable request.

REFERENCES:
- [Background] Zachovajeviene B, Siupsinskas L, Zachovajevas P, Venclovas Z, Milonas D. Effect of diaphragm and abdominal muscle training on pelvic floor strength and endurance: results of a prospective randomized trial. Sci Rep. 2019 Dec 16;9(1):19192. doi: 10.1038/s41598-019-55724-4. PMID 31844133
- [Background] Kobesova A, Davidek P, Morris CE, Andel R, Maxwell M, Oplatkova L, Safarova M, Kumagai K, Kolar P. Functional postural-stabilization tests according to Dynamic Neuromuscular Stabilization approach: Proposal of novel examination protocol. J Bodyw Mov Ther. 2020 Jul;24(3):84-95. doi: 10.1016/j.jbmt.2020.01.009. Epub 2020 Feb 8. PMID 32826013